CLINICAL TRIAL: NCT00043563
Title: Cognitive Behavioral Treatment of Pediatric Trichotillomania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21MH061457 (NIH); R21MH061457 (NIH); DSIR CT-S
Record Dates: First submitted 2002-08-09; First posted 2002-08-12 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Trichotillomania
Keywords: Cognitive-behavior Therapy; Minimal Attention Control
MeSH Terms: conditions — Trichotillomania | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Cognitive-Behavior Therapy

SUMMARY:
This study will compare the effectiveness of cognitive-behavior therapy (CBT) to a minimal attention control (AC) condition for treatment of pediatric trichotillomania (TTM).

DETAILED DESCRIPTION:
TTM is a persistent impulse control disorder in which the individual acts on urges to pull out his or her own hair. Onset typically occurs by adolescence, and TTM is often associated with significant functional impairment and distress. CBT is a type of psychotherapy designed to change problematic behaviors and thinking. It includes self-monitoring of hair-pulling urges and homework assignments to practice the use of cognitive and behavioral strategies.

Participants are assigned randomly to receive either CBT or AC for 8 weeks. Participants assigned to CBT receive weekly 1-hour sessions of CBT for 8 weeks; participants assigned to AC receive 6 telephone contacts and 2 in-person sessions for 8 weeks. After 8 weeks, CBT participants who respond to treatment enter Phase II, which lasts an additional 8 weeks and includes 4 in-person maintenance sessions. AC participants who are still symptomatic after 8 weeks are offered CBT.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Trichotillomania
* Minimum symptom duration of 6 months
* Presence of a stable parent or guardian

Exclusion Criteria:

* Other primary psychiatric diagnosis
* Bipolar illness, pervasive developmental disorder, thought disorder, current major depression, ADD/ADHD
* Concurrent psychotherapy
* Currently receiving psychotropic medications

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2001-01; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
National Institute of Mental Health (NIMH) Trichotillomania Severity Scale | 1 week
  Semi-structured interview about hair-pulling and related symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Center for the Treatment and Study of Anxiety, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Franklin ME, Edson AL, Ledley DA, Cahill SP. Behavior therapy for pediatric trichotillomania: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2011 Aug;50(8):763-71. doi: 10.1016/j.jaac.2011.05.009. Epub 2011 Jul 1. PMID 21784296
- [Derived] Franklin ME, Edson AL, Freeman JB. Behavior therapy for pediatric trichotillomania: Exploring the effects of age on treatment outcome. Child Adolesc Psychiatry Ment Health. 2010 Jun 28;4:18. doi: 10.1186/1753-2000-4-18. PMID 20584275